CLINICAL TRIAL: NCT05968573
Title: Evaluation of a Persuasive Health Communication Intervention Designed to Increase HIV/HCV Screening Among Emergency Departments Patients Who Currently, Formerly or Never Injected Drugs.
Brief Title: Persuasive Health Communication Intervention for HIV/HCV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Roland Merchant, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY-22-01162; 1R01DA055533-01 (NIH)
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Human Immunodeficiency Virus (HIV); Hepatitis C (HCV)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis C

STUDY DESIGN:
Intervention Model Description: This study has two parts:
  Part A: Modification of the PHCI with the assistance of current and former people who inject drugs (PWID) ED patients.
  Part B: Randomized Controlled Trial - this will only be conducted after completion of Part A.
Masking Description: Participants will be told during consent that they will be randomized and assigned to a group. Participants will be told that the two groups are to watch a video or listen to a health educator. Therefore, participants are not prevented from having knowledge of the interventions assigned to them.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Persuasive Health Communication Intervention delivered in video format with captions (Active Comparator): A video with captions created by the research team will be played to persuade patients to participate in HIV and Hepatitis C (HCV) screening.
  Interventions: Other: Video Format with Captions
- Persuasive Health Communication Intervention delivered in video format without captions (Active Comparator): A video with captions created by the research team will be played to persuade patients to participate in HIV and Hepatitis C (HCV) screening.
  Interventions: Other: Video Format without Captions
- Persuasive Health Communication Intervention delivered by Health Educator (Active Comparator): Healthcare provider educator getting patients screened for HIV/HCV.
  Interventions: Other: Health Educator

INTERVENTIONS:
Other: Video Format with Captions — A video with captions created by the research team will be played to persuade patients to participate in HIV and Hepatitis C (HCV) screening.
  Arms: Persuasive Health Communication Intervention delivered in video format with captions
Other: Video Format without Captions — A video without captions created by the research team will be played to persuade patients to participate in HIV and Hepatitis C (HCV) screening.
  Arms: Persuasive Health Communication Intervention delivered in video format without captions
Other: Health Educator — The video created by the research will be compared to a healthcare provider in terms of effectiveness in getting patients screened for HIV/HCV.
  Arms: Persuasive Health Communication Intervention delivered by Health Educator

SUMMARY:
A major impediment to emergency department (ED)-based HIV/HCV screening success is that often ED patients at risk for, or later diagnosed with, HIV and HCV decline testing. In this R01 project, the research team will assess how well a promising, easy-to-use, one-time, minimal-training-needed, very brief persuasive health communication intervention (PHCI) increases acceptance of testing among adult ED patients who either currently, formerly or never injected drugs and initially declined HIV/HCV screening. The research team will conduct a randomized, controlled trial (RCT) at EDs within the Mount Sinai Health System to compare the efficacy of the PHCI when delivered by a video vs. an HIV/HCV counselor. Patients who initially declined HIV/HCV screening will be stratified by injection-drug use (IDU) history cohorts: (1) current/former PWIDs, (2) never/non-PWIDs. Within each IDU history cohort, the research team will randomly assign participants (1:1:1) to a PHCI delivered by: (1) a video with captions, (2) a video without captions, (3) an HIV/HCV counselor. This R01 project will be conducted at Mount Sinai affiliate hospitals EDs. For Aim 2, the research team will determine if screening acceptance is similar across IDU history cohorts. For Aim 3, the research team will further compare the two delivery forms of the PHCI through a health economics assessment, both independent of IDU history and within each IDU history cohort.

DETAILED DESCRIPTION:
As part of routine practice at Mount Sinai Health System EDs, the ED Nurses initiate HIV/HCV screening for all patients able to provide consent. ED patients eligible for recruitment into the RCT portion of the study are those who declined HIV/HCV screening. RCs will review the electronic health records (EHRs) of patients present in the ED during data collection periods and determine which patients are potentially eligible.

Participation in the RCT involves a one-time encounter. All research-related activities will occur in the ED. As such, drop-out during this brief RCT (<30 minutes from recruitment through final study questionnaires) is expected to be minimal (<5%). RCs will coordinate with participants and ED staff to facilitate participant involvement while they are receiving medical care. If necessary, participants can continue participating in designated areas of the ED (e.g., waiting room, family room) after they are discharged and there are study-related tasks remaining. There are no research related follow-ups needed.

The research team will enroll a total of 2,000 adult ED patients who meet all study criteria and agree to participate in the RCT, stratified by IDU history. Assuming 0.6 participants completing the study/hour (1 study completion/75 minutes of recruitment, enrollment, and data collection), the research team could recruit up to ≈5,184 participants (720 collection days x 12 hours/data collection/day x 0.6 participants/hour) over 3 years.

The research team will be collecting data using the QDS™ (NOVA Research Company) program installed on a tablet computer. The program has the ability to encrypt collected data, to which only the researcher has ability to de-crypt data sets (NOVA Research cannot recover lost passwords for the researcher). The program also has a data management system, allowing data export for use in analytical packages like SPSS, Stata. Internet access is not necessary for this program to function. The data can be stored on the tablet computer for the meantime, then synced once internet is available.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years-old
* Speak English or Spanish, and able to provide informed consent for study participation
* Not HIV AND HCV infected/Antibody+ (per EHR review and patient report)
* Not already participating in a HIV or HCV study (e.g., HIV PrEP, HIV vaccine)
* Not tested for HIV OR HCV within the past 12 months (per EHR review and patient report)

Exclusion Criteria:

* <18 years old
* Unable to speak Spanish or English
* HIV or HCV positive
* Currently enrolled in another HIV or HCV research study
* Has tested for HIV or HCV in the past 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients who accept HIV/HCV testing after watching the video with captions | Day 1, up to 5 minutes after intervention
  The number of patients who accept HIV/HCV testing after watching the video with captions
Number of patients who accept HIV/HCV testing after watching the video without captions | Day 1, up to 5 minutes after intervention
  The number of patients who accept HIV/HCV testing after watching the video captions
Number of patients who accept HIV/HCV testing after speaking with a health educator | Day 1, up to 5 minutes after intervention
  The number of patients who accept HIV/HCV testing after speaking with a health educator.

SECONDARY OUTCOMES:
The number of patients that accept HIV/HCV testing by no prior injection-drug use | Day 1, up to 5 minutes after intervention
  The number of patients that accept HIV/HCV testing by no prior injection-drug use
The number of patients that accept HIV/HCV testing by former injection-drug use | Day 1, up to 5 minutes after intervention
  The number of patients that accept HIV/HCV testing by former injection-drug use
The number of patients that accept HIV/HCV testing by current injection-drug use | Day 1, up to 5 minutes after intervention
  The number of patients that accept HIV/HCV testing by current injection-drug use
Health economics assessment of PHCI | End of study, at 5 years
  The research team will further compare the two delivery forms of the PHCI through a health economics assessment, both independent of IDU history and within each IDU history cohort. This will measure cost-benefit analysis in terms of cost of each intervention in relation to how effective it is on persuading real world populations to test for HIV and HCV.

CONTACTS AND LOCATIONS:
Overall Officials: Roland C Merchant, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Specify Other Time FrameAfter last patient enrolled up to a year from that time point.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  To achieve aims in the approved proposal. Specify Other Mechanism Secured excel file sent through email.

REFERENCES:
- [Derived] Merchant RC, Harrington N, Clark MA, Liu T, Morgan J, Cowan E, Solnick R, Wyler B. Testing a persuasive health communication intervention (PHCI) for emergency department patients who declined rapid HIV/HCV screening: a randomised controlled trial study protocol. BMJ Open. 2024 Aug 12;14(8):e089265. doi: 10.1136/bmjopen-2024-089265. PMID 39134444